CLINICAL TRIAL: NCT04879914
Title: Inflammation and Intestinal Microbiota Modulation in Inflammatory Bowel Diseases
Brief Title: Analysis of Microbiota Changes Induced by Microencapsulated Sodium Butyrate in Patients With Inflammatory Bowel Disease
Acronym: IBDMicro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4049/AO/17
Record Dates: First submitted 2021-04-27; First posted 2021-05-10 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2021-09

CONDITIONS: Inflammatory Bowel Diseases; Irritable Bowel Syndrome
Keywords: IBD; Microbiota; Butyrate; IBS
MeSH Terms: conditions — Inflammatory Bowel Diseases; Irritable Bowel Syndrome | interventions — Butyrates; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butyrate (Experimental): Patients taking butyrate
  Interventions: Dietary Supplement: Butyrate
- Placebo (Experimental): Patients taking placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Butyrate — 3 cps/die 300 mg/cps
  Other Names: Butyrose
  Arms: Butyrate
Dietary Supplement: Placebo — 3 cps/die 300 mg/cps
  Other Names: starch
  Arms: Placebo

SUMMARY:
Inflammatory bowel disease (IBD) is characterized by severe inflammation of the small bowel and/or the colon leading to recurrent diarrhea and abdominal pain.

Irritable Bowel Syndrome with diarrhea (IBS-D) is characterized by abdominal pain or discomfort, gas, loose and frequent stools.

Butyrate has shown anti-inflammatory and regenerative properties, providing symptomatic relief when orally supplemented in patients suffering from various colonic diseases. The investigator proposes to investigate the effect of a microencapsulated form of sodium butyrate on the fecal microbiota of patients with IBD and IBS-D.

DETAILED DESCRIPTION:
The IBDMicro is an interventional, randomized, double-blind, placebo-controlled study. A novel oral formulation of butyrate contained in a lipophilic microcapsule, that provides extensive capacity for intestinal diffusion and facilitates slow release of the active ingredient will be used ("Butyrose" produced by SILA SRL, Italy). A proof-of-concept study has been already published in this context, and preliminary data showed that butyrate administration was able to change the gut microbiota of patients with IBD and IBS-D after 12 weeks of treatment, in association with the changes of intestinal inflammation indexes (fecal calprotectin). In keeping, investigators will assess the microbiota before and after the butyrate administration. Also, clinical data will be collected by using validated disease-specific questionnaires (Rome IV and clinical indexes for IBD). Quality of life will be also recorded. The analysis of intestinal microbiota will be carried out by collecting a fecal sample and analyzed with metagenomics techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of Crohn disease (CD) or Ulcerative colitis (UC) in the last 6 months and undergoing followup colonoscopy.

Exclusion Criteria:

* (a) prior proctocolectomy;
* (b) presence of IBD extraintestinal manifestation;
* (c) treatment with antibiotics in the last 60 days;
* (d) extensive surgical resection;
* (e) presence of stoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
NGS analysis ( 16S rRNA) will be used to highlight the microbiota variation induced by Butyrose/Placebo administration in 160 IBD and 40 IBS-D patients after 8 weeks of treatment. | 90 days
  The 16S rRNA is a fundamental component of the prokaryotic ribosome, where defines structural and functional properties interacting for example with the mRNA. Its structure and sequences were characterized during the 70's/80's, and the corresponding DNA coding sequence is referred to 16s rRNA gene. The 16s rRNA gene started to be used as the phylogenetic marker in the 70's due to its ubiquity among bacterial kingdom, allowing comparison between evolutionarily distant organisms.
  A new oral formulation of sodium-butyrate, at the dose of 3 capsules/d (1800 mg/d), will be administered, during the main meals, in consecutive IBD or IBS-D patients, for 90 days. At the same time, a control group will receive three starch capsules with similar color, flavor, and size.

SECONDARY OUTCOMES:
Treatment effects on clinical activity by fecal calprotectin. | 90 days
  Analysis of fecal calprotectin will be evaluated by clinical routinary analysis before and after treatment with Butyrose/Placebo. The Butyrose treatment at the dose of 3 capsules/die, will be administered in consecutive IBD and IBS-D patients, for 90 days. At the same time, a control group received three starch capsules with similar color, flavor, and size.
Treatment effects on lifestyle by IBD Questionaire. | 90 days
  The IBD questionnaire is a disease-specific questionnaire to highlight the patients' lifestyle before and after treatment. The IBDQ analysis will be performed as described in Yarlas A. et al.;J Patient Cent Res Rev 2020 10.17294/2330-0698.1722

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo V. Savarino, Prof. MD, PhD, Principal Investigator — Department of Surgery, Oncology and Gastroenterology - DiSCOG University of Padua - Azienza Ospedaliera di Padova
Locations (1):
- Edoardo Vinvenzo Savarino, Padua, Italy

REFERENCES:
- [Result] Facchin S, Vitulo N, Calgaro M, Buda A, Romualdi C, Pohl D, Perini B, Lorenzon G, Marinelli C, D'Inca R, Sturniolo GC, Savarino EV. Microbiota changes induced by microencapsulated sodium butyrate in patients with inflammatory bowel disease. Neurogastroenterol Motil. 2020 Oct;32(10):e13914. doi: 10.1111/nmo.13914. Epub 2020 May 31. PMID 32476236
- [Derived] Facchin S, Calgaro M, Pandolfo M, Buda A, Barberio B, Zingone F, Vitulo N, Savarino EV. Impact of oral butyrate on clinical and biochemical parameters in IBD: A randomized placebo-controlled study targeting gut microbiota. Dig Liver Dis. 2026 Jan;58(1):64-73. doi: 10.1016/j.dld.2025.11.014. Epub 2025 Dec 6. PMID 41354580